CLINICAL TRIAL: NCT04369495
Title: BAFF Levels After Cyclophosphamide and Mycophenolate Use in Patients With Systemic Lupus Erythematosus
Brief Title: BAFF Levels and Lupus Nephritis (LN)
Acronym: BAFF
Status: Withdrawn | Type: Observational
Why Stopped: Legal problems with financial support, The study never began
Sponsor: Universidad de Antioquia (Other)
Collaborators: ARTMEDICA (Unknown)
Responsible Party: Principal Investigator, Gloria Vasquez, MD, DrSc, Rheumatologyst, Prinicipal investigator, Proffesor Grupo de Inmunologia Celular e Inmunogenética. Instituto de Investigaciones Médicas. Facultad de Medicina., Universidad de Antioquia
Other Study IDs: UAntioquia/GICIG/BAFF
Record Dates: First submitted 2020-04-27; First posted 2020-04-30 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Lupus Nephritis
Keywords: BAFF
MeSH Terms: conditions — Lupus Nephritis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cyclophosphamide: Patients with induction therapy for lupus nephritis with cyclophosphamide
  Interventions: Other: BAFF serum levels
- Mycophenolate: Patients with induction therapy for lupus nephritis with mycophenolate
  Interventions: Other: BAFF serum levels

INTERVENTIONS:
Other: BAFF serum levels — BAFF levels in serum in visit 0,1,2 during induction therapy

SUMMARY:
B-cell activating factor (BAFF), serves as a vital survival and differentiation factor for normal B-cell development. BAFF levels have been associated with the clinical activity of SLE in humans. BAFF plays a pathogenic role in SLE in part through T cell-dependent B cell autoantibody production. BAFF, has a role in the maintenance of memory B cells and promotes plasma cell survival. Treatment strategies involving BAFF blockade haven been studied in patients with SLE inducing overall improvement in disease activity, mainly in musculoskeletal and mucocutaneous domains leading to the approval of Belimumab for the treatment of patients with SLE without severe renal or neurological involvement.

Antibodies against CD20 molecule, (Rituximab), cyclophosphamide (CYC), and mycophenolate (MMF) have all been used for the treatment of different manifestations of SLE and both moderate and severe activity. Baseline C4 level, early normalization of complement, and reduction in proteinuria have been shown to predict renal response to therapy with MMF or CYC in lupus nephritis. With Rituximab (RTX), B cell depletion has been associated with response to treatment and relapse prediction. The elevation of serum BAFF levels after B cell depletion with RTX in SLE are associated with anti-double-stranded DNA antibody levels and disease flare. The rise of BAFF is probably due to the decrease in its receptors leading to a release of BAFF and a delayed regulation of BAFF mRNA transcription, both of which could favor the re-emergence of autoreactive B cells. It has been suggested that the rise in BAFF levels after anti-CD20 therapy might be related to flares of the disease. Additionally, the combination of anti-CD20 with anti-BAFF or antibodies against CD4, reduces the number of splenic plasma cells in mouse models and has been proven to have a lasting benefit both in lupus-prone mice and in mice with established disease. Currently, there is a lack of information regarding MMF or CYC and BAFF levels. We consider that it is fundamental to know the behavior of BAFF in patients with SLE after treatment with MMF or CYC bearing in mind the proposal of multiple experts of the possible use of sequential therapy of BAFF inhibition after B-cell depletion. Knowledge of the behavior of BAFF will allow me to better understand its implications in SLE and its therapy and postulate the use of sequence therapy with Belimumab after CYC o MF induction with the proposal to reduce the flares

DETAILED DESCRIPTION:
1.3. Research question Flares of lupus nephritis are related to the behavior of BAFF levels before, during, and after induction therapy.

2. Theoretical framework B-cell activating factor (BAFF), also known as B lymphocyte stimulator (BLyS) serves as a vital survival and differentiation factor for normal B-cell development. There is an inverse relationship between BAFF circulating levels and the percentage and number of circulating B cells. APRIL (a proliferation-inducing ligand) shares substantial homology with BAFF and binds to two of the three BAFF receptors (BCMA and TACI) but not to BR3. Like BAFF, APRIL has little role in the maintenance of memory B cells but does promote plasma cell survival better than does BAFF. Both BAFF and APRIL levels behave differently after B cell depletion in SLE and rheumatoid arthritis. BAFF levels have been associated with the development of systemic lupus erythematosus (SLE) in murine models and with clinical activity of SLE in humans. BAFF plays a pathogenic role in SLE in part through T cell-dependent B cell autoantibody production. Treatment strategies involving BAFF blockade haven been studied in patients with SLE inducing overall improvement in disease activity, mainly in musculoskeletal and mucocutaneous domains leading to the approval of Belimumab for the treatment of patients with systemic lupus erythematosus without severe renal or neurological involvement.

Anti-CD20 antibodies (Rituximab), cyclophosphamide (CYC), and mycophenolate (MMF) have all been used for the treatment of systemic lupus erythematosus, and both moderate and severe activity. Both MMF and CYC show a significant effect on disease activity and circulating B, T, Natural Killer cells (NK), and Natural Killer T cells (NKT) cell subsets. Baseline C4 level, early normalization of complement, and reduction in proteinuria have been shown to predict renal response to therapy with MMF or CYC in lupus nephritis. With Rituximab (RTX), B cell depletion has been associated with response to treatment and relapses. The elevation of serum BAFF levels after B cell depletion with RTX in SLE are associated with anti-double-stranded DNA antibody levels and disease flare. The rise of BAFF is probably due to the decrease in its receptors leading to a release of BAFF and a delayed regulation of BAFF messenger-RNA (mRNA) transcription, both of which could favor the re-emergence of autoreactive B cells.

It has been suggested that the rise in BAFF levels after anti-CD20 therapy might be related to flares of the disease and that repeated rituximab infusions can result in a feedback loop characterized by ever-rising BAFF levels, surges in autoantibody production and worsening of the disease. Additionally, the combination of antiCD20 with anti-BAFF or anti-CD4 antibody greatly reduces the number of splenic plasma cells in mouse models and anti-CD20 plus anti-BAFF has been proven to have a lasting benefit both in lupus-prone mice and in mice with established disease.

B-cell depletion therapy (BCDT) has been used in patients with refractory disease with failure to standard therapy through a combination of RTX and CYC, which showed an improvement in clinical and serological disease activity. Serological findings suggest that B cell clones committed to producing antinucleosome antibodies and anti-dsDNA have a relatively rapid turnover compared with cell clones producing other autoantibodies(30). BAFF levels rose in most patients at 3 months post BCDT. Those patients with an expanded autoantibody profile and raised BAFF levels at baseline had shorter responses to BCDT. Retreatment with BCDT may produce a more sustained clinical response.

Currently, there is a lack of information regarding MMF or CYC and BAFF levels without the use of concomitant RTX (for CYC) and in monotherapy (for MMF). We consider that it is fundamental to know the behavior of BAFF in patients with SLE after treatment with MMF or CYC bearing in mind the proposal of multiple experts of the possible use of sequential therapy of BAFF inhibition after B-cell depletion. Knowledge of the behavior of BAFF will allow to better understand its implications in SLE and its therapy.

3. Hypothesis Elevated BAFF levels after induction therapy with MMF or CYC is associated with disease relapse.

4. Objectives 4.1. Main objective Analyze the relationship between BAFF levels and relapses after treatment with CYC and MMF

4.2. Specific objectives

* Describe the clinical and immuno-serological characteristics of patients with lupus nephritis at weeks 0, 12, and 24 of induction therapy.
* Compare the effects of CYC and MMF on BAFF levels in patients with lupus nephritis in induction therapy
* Evaluate the association between BAFF levels and remission of lupus nephritis treated with CYC and MMF.

ELIGIBILITY:
Inclusion Criteria:

1. Patients are older than 18 years
2. Patients that fulfill any of the available classification criteria for systemic lupus erythematosus
3. Patients with new-onset lupus nephritis or with lupus nephritis relapse after successful remission.
4. Patients with a diagnosis of lupus nephritis according to Wallace and Dubois criteria
5. Patients with class III and IV lupus nephritis with or without Class V lupus nephritis.

Exclusion Criteria:

1. Women with a positive pregnancy test
2. Class I, II, V lupus nephritis without Class III or IV lupus nephritis
3. Patients with an active malignancy or active treatment for malignancy.
4. Patients with kidney disease with GFR <30ml / min
5. Patients with severe leukopenia
6. Patients with active infection

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Patients with SLE diagnosis that fulfill either the 1987 American College of Rheumatology Classification Criteria for SLE, 2011 Systemic Lupus International Collaborating Clinics (SLICC) classification criteria for systemic lupus erythematosus or 2019 EULAR/ACR Lupus Classification criteria.
  * There will not be a successive recruitment of patients. Instead, there will be a deliberate recruitment aiming to maintain the proportion of patients needed for each group.
  A sample will be taken for the convenience of 30 patients with lupus nephritis by Wallace and Dubois criteria. Fifteen patients under treatment with CYC and 15 patients treated with MMF are selected according to the decision of the attending physician.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-01 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Levels of BAFF | Time 0, beginning of the induction therapy
  Levels of BAFF
Levels of BAFF | Time 1, 12 weeks after beginning of induction therapy
  Levels of BAFF
Levels of BAFF | Time 2, 24 weeks after beginning of induction therapy
  Levels of BAFF
Lupus Clinical Manifestations | Time 0, beginning of the induction therapy
  All clinical manifestations associated with SLE
Lupus Clinical Manifestations | Time 1, 12 weeks after beginning of induction therapy
  All clinical manifestations associated with SLE
Lupus Clinical Manifestations | Time 2, 24 weeks after beginning of induction therapy
  All clinical manifestations associated with SLE
Serological findings | Time 0, beginning of the induction therapy
  Serological parameters evaluated including anti-DNA
Serological findings | Time 1, 12 weeks after beginning of induction therapy
  Serological parameters evaluated including anti-DNA
Serological findings | Time 2, 24 weeks after beginning of induction therapy
  Serological parameters evaluated including anti-DNA
Inflammatory cytokine levels | Time 0, beginning of the induction therapy
  Cytokine levels IL-10, IL-12, TNF-α, IL-1β, IL-8 e IL-6
Inflammatory cytokine levels | Time 1, 12 weeks after beginning of induction therapy
  Cytokine levels IL-10, IL-12, TNF-α, IL-1β, IL-8 e IL-6
Inflammatory cytokine levels | Time 2, 24 weeks after beginning of induction therapy
  Cytokine levels IL-10, IL-12, TNF-α, IL-1β, IL-8 e IL-6

CONTACTS AND LOCATIONS:
Overall Officials: Gloria Vasquez, MD, DrSc, Principal Investigator — Universidad de Antioquia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schneider P, MacKay F, Steiner V, Hofmann K, Bodmer JL, Holler N, Ambrose C, Lawton P, Bixler S, Acha-Orbea H, Valmori D, Romero P, Werner-Favre C, Zubler RH, Browning JL, Tschopp J. BAFF, a novel ligand of the tumor necrosis factor family, stimulates B cell growth. J Exp Med. 1999 Jun 7;189(11):1747-56. doi: 10.1084/jem.189.11.1747. PMID 10359578
- [Background] Kreuzaler M, Rauch M, Salzer U, Birmelin J, Rizzi M, Grimbacher B, Plebani A, Lougaris V, Quinti I, Thon V, Litzman J, Schlesier M, Warnatz K, Thiel J, Rolink AG, Eibel H. Soluble BAFF levels inversely correlate with peripheral B cell numbers and the expression of BAFF receptors. J Immunol. 2012 Jan 1;188(1):497-503. doi: 10.4049/jimmunol.1102321. Epub 2011 Nov 28. PMID 22124120
- [Background] Petri M, Stohl W, Chatham W, McCune WJ, Chevrier M, Ryel J, Recta V, Zhong J, Freimuth W. Association of plasma B lymphocyte stimulator levels and disease activity in systemic lupus erythematosus. Arthritis Rheum. 2008 Aug;58(8):2453-9. doi: 10.1002/art.23678. PMID 18668552
- [Background] Salazar-Camarena DC, Ortiz-Lazareno PC, Cruz A, Oregon-Romero E, Machado-Contreras JR, Munoz-Valle JF, Orozco-Lopez M, Marin-Rosales M, Palafox-Sanchez CA. Association of BAFF, APRIL serum levels, BAFF-R, TACI and BCMA expression on peripheral B-cell subsets with clinical manifestations in systemic lupus erythematosus. Lupus. 2016 May;25(6):582-92. doi: 10.1177/0961203315608254. Epub 2015 Sep 29. PMID 26424128
- [Background] Vallerskog T, Heimburger M, Gunnarsson I, Zhou W, Wahren-Herlenius M, Trollmo C, Malmstrom V. Differential effects on BAFF and APRIL levels in rituximab-treated patients with systemic lupus erythematosus and rheumatoid arthritis. Arthritis Res Ther. 2006;8(6):R167. doi: 10.1186/ar2076. PMID 17092341
- [Background] Manzi S, Sanchez-Guerrero J, Merrill JT, Furie R, Gladman D, Navarra SV, Ginzler EM, D'Cruz DP, Doria A, Cooper S, Zhong ZJ, Hough D, Freimuth W, Petri MA; BLISS-52 and BLISS-76 Study Groups. Effects of belimumab, a B lymphocyte stimulator-specific inhibitor, on disease activity across multiple organ domains in patients with systemic lupus erythematosus: combined results from two phase III trials. Ann Rheum Dis. 2012 Nov;71(11):1833-8. doi: 10.1136/annrheumdis-2011-200831. Epub 2012 May 1. PMID 22550315
- [Background] Moroni G, Raffiotta F, Trezzi B, Giglio E, Mezzina N, Del Papa N, Meroni P, Messa P, Sinico AR. Rituximab vs mycophenolate and vs cyclophosphamide pulses for induction therapy of active lupus nephritis: a clinical observational study. Rheumatology (Oxford). 2014 Sep;53(9):1570-7. doi: 10.1093/rheumatology/ket462. Epub 2014 Feb 6. PMID 24505125
- [Background] Fassbinder T, Saunders U, Mickholz E, Jung E, Becker H, Schluter B, Jacobi AM. Differential effects of cyclophosphamide and mycophenolate mofetil on cellular and serological parameters in patients with systemic lupus erythematosus. Arthritis Res Ther. 2015 Apr 3;17(1):92. doi: 10.1186/s13075-015-0603-8. PMID 25890338
- [Background] Zhao L, Jiang Z, Jiang Y, Ma N, Wang K, Zhang Y. Changes in immune cell frequencies after cyclophosphamide or mycophenolate mofetil treatments in patients with systemic lupus erythematosus. Clin Rheumatol. 2012 Jun;31(6):951-9. doi: 10.1007/s10067-012-1958-8. Epub 2012 Feb 21. PMID 22349930